CLINICAL TRIAL: NCT02995226
Title: Analysis of the Capacity to Regulate Physical Efforts and to Estimate Its Intensity as an Endophenotype of Anorexia Nervosa, Because of a Specific Impact of the Physical Effort at the Emotional, Cognitive, Pain, Genetic and Biological Level
Brief Title: Abnormal Regulation, Estimation and Cognitive Impacts of Physical Efforts as an Endophenotype of Anorexia Nervosa
Acronym: CAPANOX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: D15-P018
Record Dates: First submitted 2016-12-05; First posted 2016-12-16 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa | interventions — Surveys and Questionnaires; Restraint, Physical; Blood Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anorexia nervosa (Other): Patients with DSM-5 criteria of "anorexia nervosa"
  Interventions: Other: Clinical and biological examination, Saliva (or blood) test Glycemia, thermal test, cognitive and bike tests, questionnaires
- First degree relatives (Other): First degree relatives (of patients suffering from anorexia nervosa) with no eating disorder
  Interventions: Other: Clinical examination, Glycemia, saliva (or blood) test, thermal test, cognitive and bike tests, questionnaires
- Controls (with no eating disorder) (Other): Other
  Interventions: Other: Clinical examination, Glycemia, saliva (or blood) test, thermal test, cognitive and bike tests, questionnaires

INTERVENTIONS:
Other: Clinical and biological examination, Saliva (or blood) test Glycemia, thermal test, cognitive and bike tests, questionnaires — Clinical and biological examination, Saliva (or blood) test, glycemia, thermal test, cognitive and bike tests, questionnaires
  Arms: Anorexia nervosa
Other: Clinical examination, Glycemia, saliva (or blood) test, thermal test, cognitive and bike tests, questionnaires — Clinical examination, Glycemia, saliva (or blood) test, thermal test, cognitive and bike tests, questionnaires
  Arms: Controls (with no eating disorder); First degree relatives

SUMMARY:
The purpose of this study is to check if patients, but also relatives (as they share familial and genetic risk factors), are having more difficulties in regulating a spontaneous, pleasant physical effort (doing "too much") compared to healthy controls, and if physical efforts are participating to core symptoms of anorexia nervosa, such as more appetite (instead of less), less pain, more abnormal body image, and less cognitive flexibility.

Such a result could help to further understand the role of difficulties with physical exercise as part of the phenotype of anorexia nervosa.

DETAILED DESCRIPTION:
This is a three steps protocol. First, patients (with anorexia nervosa), controls (with no eating disorder) and first degree relatives (with no eating disorder) will be tested for emotional accuracy (seing faces on a screen with different core emotions), pain threshold (how long they can support a cold probe), body size (how they see themselves), appetite and cognitive flexibility (a test where the capacity to change rules during a game is done easily or not).

Then all subjects will do a standardized physical exercise which represents an effort with the equivalent level of energy for each participants as being chosen according to each level of competency (assessed through the "maximal aerobic power").

The third step consists in the repetition of (nearly) initial tests.

ELIGIBILITY:
Inclusion Criteria:

Patients :

* Woman
* 18 - 50 years
* eating disorders (with or without bulimia) according to the EDI-2 (Eating Disorder Inventory) and the MINI (Mini International Neuropsychiatric Interview)
* BMI (Body Mass index) between 14 and 17,5
* first degree relative without ED (eating disorders)

First degree relatives :

* Woman
* 18 - 50 years
* Mother or sister of patient with eating disorders
* BMI (Body Mass index) upper to 17,5
* Healthy of all ED (eating disorders)

Controls :

* Woman
* 18 - 50 years
* BMI > 17,5
* Without ED (eating disorders)

Exclusion Criteria:

All groups :

* Contraindication in the practice of an intensive sport
* Cardiovascular Family history with risk of cardiovascular unwanted events
* Cardiovascular, surgical personal Histories, ostéoarticulaires or musculo-tendinous against indicating to the practice of a sport
* Intercurrents psychiatric pathologies (humor or psychotics disorders, chronic or acute)

Related and controls :

Diagnosis of ED (eating disorders) in the EDI-2 and in the MINI

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-02-27 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Physical power | Day 0
  Comparison inter and intra individual of the subjective and objective power to the subjects during a typical physical bike test.

SECONDARY OUTCOMES:
Pain threshold | Day 0
  This threshold is based on the minimum temperature that the patient is able to suppor (the probe is placed on the skin of the forarm, and the temperature reduces its temperature every 10 seconds), knowing that the machine is not getting to temperatures that can be damageable.
  Comparison before and after bike test
Wellbeing self-questionnaire | Day 0
  Comparison before and after bike test
Hunger Visual analogical scale | Day 0
  Comparison before and after bike test
PANAS score (self-questionnaire) | Day 0
  Emotions. Comparison before and after bike test
Hunger Visual analogical scale | Day 0
  Apetite. Comparison before and after bike test
Performance on the Briton cognitive test (number of errors) | Day 0
  Mental flexibility. Comparison before and after bike test
Performance on cognitive tests (speed, number of errors), before versus after the exercise, in the three groups. | Day 0
  Tests. Performance on cognitive tests (speed, number of errors), before versus after the exercise, in the three groups.
Genetical analysis | Day 0
  10 candidate genes will be analyzed (following the collection of blood or saliva) assessing the frequency of their main alleles (variants), looking for a significant difference of allele frequency between the 3 groups.

CONTACTS AND LOCATIONS:
Overall Officials: Philip GORWOOD, MD, PhD, Study Chair — CHSA
Locations (1):
- Centre Hospitalier Sainte Anne, Paris, France

IPD SHARING:
Plan to Share IPD: No